CLINICAL TRIAL: NCT04240418
Title: Initiative in LYon for Lung cAncer Screening Development - Prevalence Study
Acronym: ILYAD1
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: ILYAD1_2019
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Lung Cancer; Screening
MeSH Terms: conditions — Lung Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lyon University Hospital employees
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — The objective is to evaluate the eligibility of the responders, as defined by NELSON criteria and PLCOm2012 scoring, and their willingness to participate to a lung-cancer screening with low-dose computed tomography.

SUMMARY:
Screening at-risk subjects with low-dose computed tomography (CT) efficiently reduces lung cancer specific mortality. However screening efficiency relies on the at-risk population's criteria definition and its participation rate to the screening. In France, there are concerns regarding the participation rates to national cancer screening that are quite low (around 50% and 32% of the eligible population for breast cancer and colorectal cancer respectively). Before organizing national lung cancer screening it is then crucial to determine the factors impacting the at-risk subjects willingness to participate in lung cancer screening.

The Lyon University Hospital is the second biggest hospital in France with more than 23,000 employees distributed among more than 160 professions representing every level of education or working conditions. Its population is heterogeneous and wide enough to perform a prevalence study assessing the willingness to participate among the at-risk population.

ILYAD is a prospective study performed by anonymous questionnaires that will be submitted to the 23,000 employees of the Lyon University Hospital. The study main objective is to evaluate the at-risk population presence in the Lyon University Hospital population, as defined by NELSON criteria and selection criteria for lung cancer screening (PLCOm2012 scoring), and its willingness to participate to a lung-cancer screening with low-dose CT. This might help further efficient national lung cancer screening campaign organization.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Employee from the Lyon University Hospital (receiving salary from the Lyon University Hospital)
* Person who has willingness to respond the survey

Exclusion Criteria:

* Employees not hired by the Lyon University Hospital
* Employees who have not willingness to participate in the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Civil Hospices of Lyon is the second largest university hospital in France, with 23000 staff.
Sampling Method: Non-Probability Sample
Enrollment: 4595 (Actual)
Dates: Start 2020-10-31 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Number of employees belonging to the at-risk population for lung cancer and consequently eligible to lung cancer screening. | Day 0 (at inclusion)
  High-risk ever-smokers are defined as ever-smokers aged 55-74 years old, having smoked >15 cigarettes per day for >25 years or >10 cigarettes for >30 years and with ≤15 years since cessation for quitters.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France